CLINICAL TRIAL: NCT05678933
Title: Phase 3 Multi-center Randomized Study to Compare Efficacy and Safety of Azacitidine and Chidamide Combined With CHOP (AC-CHOP) Versus CHOP in Patients With Previously Untreated Peripheral T-cell Lymphoma With T-follicular Helper Phenotype (PTCL-TFH)
Brief Title: AC-CHOP Versus CHOP in Patients With Previously Untreated PTCL-TFH
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Principal Investigator, Huilai Zhang, Chief of department of lymohoma, Tianjin Medical University Cancer Institute and Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AC-CHOP Study
Record Dates: First submitted 2022-12-28; First posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Peripheral T-cell Lymphoma Targeted Therapy
MeSH Terms: interventions — Azacitidine; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Cyclophosphamide; Epirubicin; Vincristine; Prednisone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AC-CHOP (Experimental): Azacitidine administered IV at day 1-5 and Chidamide admistered twice a week for two weeks in combination with cyclophosphamide, doxorubicin, vincristine and prednisone (CHOP)
  Interventions: Drug: Azacitidine; Drug: Chidamide; Drug: Cyclophosphamide; Drug: Epirubicin; Drug: Vincristine; Drug: Prednisone
- CHOP (Active Comparator): CHOP administered every 3 weeks for 6 cycles.
  Interventions: Drug: Cyclophosphamide; Drug: Epirubicin; Drug: Vincristine; Drug: Prednisone

INTERVENTIONS:
Drug: Azacitidine — Azacitidine (75mg/ m2) will be administered at day 1-5 by subcutaneous injection of each 21-day cycle.
  Arms: AC-CHOP
Drug: Chidamide — Chidamide (20 mg) will be taken orally twice a week for two weeks of each 21-day cycle.
  Arms: AC-CHOP
Drug: Cyclophosphamide — Cyclophosphamide (750 mg/ m2) will be administered by an intravenous infusion on day 1 of each 21-day cycle.
Drug: Epirubicin — Epirubicin (70mg/ m2) will be administered by an intravenous infusion on day 1 of each 21-day cycle.
Drug: Vincristine — Vincristine (1.4mg/ m2，Max dose 2mg) will be administered by an intravenous injection on day 1of each 21-day cycle.
Drug: Prednisone — Prednisone (100 mg) will be taken orally from day 1-5 of each 21-day cycle.

SUMMARY:
This study is an open label, multicenter study. Subjects are randomized at a 1:1 ratio to receive either (arm A) azacitidine administered IH at day 1-5 and chidamide admistered twice a week for two weeks in combination with cyclophosphamide, doxorubicin, vincristine and prednisone (CHOP) or (arm B) CHOP administered every 3 weeks for 6 cycles in patients with previously untreated peripheral T-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

Patients must satisfy all following criteria to be enrolled in the study:

1. Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures are conducted.
2. Males and females of 18 years of age to 70 years of age.
3. ECOG performance status 0, 1 or 2
4. Patients with histologically proven peripheral T-cell lymphoma with T-follicular helper phenotype (PTCL-TFH); the following subtypes as defined by the WHO classification (5th) may be included, whatever the Ann Arbor stage (I - IV):

   i.Angioimmunoblastic T-cell lymphoma ii. peripheral T-cell lymphoma of follicular type iii. Nodal and extra-nodal peripheral T cell lymphoma with follicular helper T cell phenotype
5. Previously received no treatment for PTCL, including chemotherapy, targeted therapy, immunotherapy, local radiotherapy for lymphoma (except for relieving tumor-related symptoms), surgical treatment (except for tumor or pathological tissue biopsy)
6. Life expectancy of ≥ 90 days (3 months)
7. At least one evaluable or measurable lesion that meets Lugano2014 criteria: lymph node lesions, which are measurable > 1.5 cm, and non-lymph node lesions, which are measurable>1.0 cm
8. Female and males patients of child bearing potential must use an effective method of birth control (i.e. hormonal contraceptive, intrauterine device, diaphragm with spermicide, condom with spermicide or abstinence) during treatment period and 12 month thereafter
9. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L, Platelet count ≥ 80 x 109/L, Haemoglobin ≥ 90g/L
10. Serum creatinine ≤ 1.5 x upper limit of normal (ULN) , AST or ALT ≤ 2.5 x ULN (≤ 5 x ULN for liver involvement), serum total bilirubin ≤ 1.5 x ULN (≤ 3 x ULN for liver involvement)
11. Able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

Presence of any of the following will exclude a patient from enrollment:

1. Previous treatment for PTCL with immunotherapy or chemotherapy except for short-term corticosteroids (duration of ≤ 8 days) before randomization
2. Contraindication to any drug contained in the chemotherapy regimen
3. Previous or current malignancies other than lymphoma (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast have been effectively controlled) unless the patient has been free of the disease for ≥ 5 years
4. Primary or secondary central nervous system (CNS) lymphoma involvement or having a history of CNS lymphoma at the time of recruitment
5. Undergone major surgical procedures within 14 days prior to the first dose of study drug
6. Significant and uncontrolled cardiovascular disease at screening
7. Any of the following laboratory abnormalities, except if secondary to the lymphoma:

   1. Absolute neutrophil count (ANC) < 1,000 cells/mm3 (1.0 x 109/L),
   2. Platelet count < 50,000/mm3 (50 x 109/L)
   3. Serum total bilirubin > 2 x ULN, serum ALT or AST > 3.0 x upper limit of normal (ULN), except if investigator believes that the abnormal liver function is caused by the disease
   4. Serum creatinine > 2.0 x ULN, except if investigator believes that the abnormal liver function is caused by the disease
8. Uncontrolled active systemic fungal, bacterial, viral or other infections
9. Subjects with HIV positivity
10. Subjects with active hepatitis B or C (HBs Ag+/HBc Ab+ and HBV DNA>1x103copy/mL; HCV DNA>1x103copy/mL)
11. Pregnant or lactating females or women of childbearing potential not willing to use an adequate method of birth control for the duration of the study.
12. Other situations that investigators considered inappropriate for enrollment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Insititute & Hospital, Tianjin, Tianjin Municipality, China